CLINICAL TRIAL: NCT03408574
Title: The Nicotinic Cholinergic System and Cognitive Aging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Julie Dumas, Associate Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CHRMS 16-284
Record Dates: First submitted 2018-01-03; First posted 2018-01-24 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Healthy Aging
Keywords: nicotinic system; cognitive aging; working memory; fMRI
MeSH Terms: interventions — Tobacco Use Cessation Devices; Mecamylamine

STUDY DESIGN:
Intervention Model Description: Healthy older adults aged 65-75 and healthy younger adults aged 18-30 will be recruited. Each participant will take part in 3 nicotinic drug challenge days. The three drugs are counterbalanced across study days within each group and balanced by sex.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a double blind study. The PI and all study personnel are blinded. Only the pharmacist dispensing the medication and the biostatistician who created the counterbalancing order are unblended.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Older Adults (Experimental): Healthy adults aged 65-75 will participate in three study days where they are randomly assigned to receive either nicotine patch, oral mecamylamine, placebo and perform a working memory task during the fMRI. BOLD signal is the outcome measure.
  Interventions: Drug: Nicotine patch, oral mecamylamine, placebo
- Younger Adults (Experimental): Healthy adults aged 18-30 will participate in three study days where they are randomly assigned to receive either nicotine patch, oral mecamylamine, or placebo and perform a working memory task during the fMRI.BOLD signal is the outcome measure.
  Interventions: Drug: Nicotine patch, oral mecamylamine, placebo

INTERVENTIONS:
Drug: Nicotine patch, oral mecamylamine, placebo — Each participant randomly receives one active drug or placebo on each of three study days.

SUMMARY:
Prior research has shown that a chemical system in the brain called the cholinergic system is primarily responsible for cognitive symptoms seen in people with dementia. While therapeutic benefits are clear in dementia, what remains uncertain is the role that the cholinergic system in general and a subset of receptors called the nicotinic system plays in cognition in healthy non-demented older adults (referred to as normal cognitive aging). This is critical because the ever growing healthy aging population will show declines in cognition that fall short of dementia but still impact functional abilities and independence. Maintaining good nicotinic system functioning throughout adulthood may lessen the cognitive symptoms of aging. At this time, it is not clear what the biological cause of age-related changes in cognition is. This study will examine the role of the nicotinic system in the healthy aging brain and examine its role in memory and thinking processes in older and younger adults.

DETAILED DESCRIPTION:
The cholinergic system has been shown to be the primary neurotransmitter system responsible for cognitive symptoms in dementia. While therapeutic benefits are clear in dementia, what remains uncertain is the role that the cholinergic system in general and the nicotinic system specifically plays in cognition in healthy non-demented older adults (referred to as normal cognitive aging in this application). This is critical because the expansion of the healthy aging population will nonetheless show declines in cognition that fall short of dementia but still impact functional abilities and independence. Understanding the effects of age-related functional changes on the nicotinic system will elucidate one neurochemical mechanism underlying age-related changes in cognition and will provide information about how nicotinic dysfunction affects cognition in healthy older adults. Prior research has shown that the nicotinic system has a roll in attention and memory in healthy adults. More recently, with the increased use of brain functional magnetic resonance imaging (fMRI) in combination with psychopharmacological manipulations, data patterns have emerged that further define the role of the nicotinic system in cognition, aging, and dementia.

The investigators propose that nicotinic system changes are responsible for age differences in working memory task performance and brain activation. The investigators can observe the functioning of the nicotinic system by examining brain activation patterns in response to nicotinic blockade and stimulation. Increased dorsolateral prefrontal cortex (DLPFC) activation has been shown for older adults compared to younger adults and is hypothesized to be a compensation response for the aging process. The investigators propose that temporary antagonism of the nicotinic system will also produce increased DLPFC activation. However, the relationship between this increased activation and performance will be in different directions for older and younger adults. In older adults, the increased activation will be positively correlated with performance because it is a compensatory response. In younger adults, the increased activation will be negatively correlated with performance because it is a non-adaptive response to the temporary nicotinic antagonism. Nicotinic stimulation in older adults will reveal decreased DLPFC activation that will be negatively correlated with performance and this represents the "younger" pattern of the performance and activation relationship. The younger adults will have a similar pattern of activation and performance as the older adults after nicotinic stimulation because they are already performing optimally and will not receive any further enhancement. These data will further the understanding of a neurochemical mechanism involved in normal aging and how brain activation patterns relate to receptor function.

ELIGIBILITY:
Inclusion Criteria:

* Normal cognition, not demented, no mild cognitive impairment. IQ greater than 80.

Exclusion Criteria:

* Current use of barbiturates, rifampin, insulin, carbamezepine, oral hypoglycemics, antidepressants, diabetes, or untreated thyroid disease.
* In addition, the following exclusions are specific for the challenge drugs: heavy alcohol or coffee use, significant cardiovascular disease, ischemic heart disease, asthma, chronic obstructive pulmonary disease, active peptic ulcer, hyperthyroidism, pyloric stenosis, narrow angle glaucoma, epilepsy, or current Axis I psychiatric disorders.
* Current use of centrally active drugs and drugs with cholinergic properties. A minimum of 14 days will elapse between discontinuing centrally active or psychoactive agents and this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Age effects of nicotinic blockade | After the completion of the third study day.
  Examine the effects of nicotinic blockade compared to placebo on the relationship between working memory performance and brain activation using fMRI BOLD signal in older and younger adults.
Age effects of nicotinic stimulation | After the completion of the third study day.
  Examine the effects of nicotinic stimulation compared to placebo on the relationship between working memory performance and brain activation using fMRI BOLD signal in older and younger adults.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Dumas, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be available to be shared with other researchers. The Principal Investigator will make fMRI and behavioral data available as requested by researchers after the study is completed and data sets have been cleaned for quality and locked.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03408574/Prot_SAP_000.pdf